CLINICAL TRIAL: NCT02049099
Title: A Non-interventional Retrospective Study of the Current Treatment Practice in European Haemophilia Care
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.HAEM89-001
Record Dates: First submitted 2014-01-28; First posted 2014-01-29 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Haemophilia A; Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To describe the current treatment practice during 12 months for previously treated patients diagnosed with haemophilia A or haemophilia B.

DETAILED DESCRIPTION:
The study population consists of patients with a diagnosis of ICD10: haemophilia A D66.9 or haemophilia B D67.9.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with severe or moderate haemophilia A or haemophilia B.
* Treatment with Factor VIII/Factor IX products initiated at least 24 months before inclusion in the study.
* Informed consent is obtained from the patient or patient's legal representative (as applicable according to legal regulation).

Exclusion Criteria:

* Confirmed positive inhibitor test detected in the past 24 months.

Min Age: 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients with a diagnosis of ICD10: haemophilia A D66.9 or haemophilia B D67.9.
Sampling Method: Non-Probability Sample
Enrollment: 1658 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Total dose (IU) issued of Factor VIII during a 12 month period | - 12 month to Day 0
Total dose (IU) issued of Factor IX during a 12 month period | - 12 month to Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lethagen, MD, Study Director — Swedish Orphan Biovitrum AB (publ)
Locations (12):
- Swedish Orphan Biovitrum Investigational Site, Brussels, Belgium
- France (2):
  - Swedish Orphan Biovitrum Investigational Site, Montpellier
  - Swedish Orphan Biovitrum Investigational Site, Nantes
- Germany (2):
  - Swedish Orphan Biovitrum Investigational Site, Bonn
  - Swedish Orphan Biovitrum Investigational Site, Leipzig
- Italy (3):
  - Swedish Orphan Biovitrum Investigational Site, Florence
  - Swedish Orphan Biovitrum Investigational Site, Milan
  - Swedish Orphan Biovitrum Investigational Site, Vicenza
- Spain (2):
  - Swedish Orphan Biovitrum Investigational Site, Barcelona
  - Swedish Orphan Biovitrum Investigational Site, Madrid
- Swedish Orphan Biovitrum Investigational Site, Stockholm, Sweden
- UKHCDO, Manchester, United Kingdom